CLINICAL TRIAL: NCT02216734
Title: Effects of Mother Support Groups on Prevention of Mother-To-Child Transmission (PMTCT) Outcomes in Mutare & Makoni Districts, Zimbabwe: A Cluster Randomized Controlled Trial
Brief Title: Effects of Facility-based Mother Support Groups on Prevention of mother-to Child Transmission Outcomes in Zimbabwe
Acronym: EPAZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Family AIDS Caring Trust (Other)
Collaborators: World Health Organization (Other); Canadian International Development Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RPC526
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: HIV Infection
Keywords: HIV/AIDS; Prevention of mother-to-child transmission; Mother support groups; Retention-in-care; Male participation; Anti-retroviral treatment; Infants
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mother support groups for HIV+ mothers (Experimental): Facility-based mother support groups (MSGs) for HIV+ mothers. MSGs were established prior to study enrolment. MSGs are facilitated by volunteer mothers. Groups meet every two weeks. Health information is provided by health workers during MSGs. Mothers receive HIV prevention, psychosocial and treatment support, reinforce safe feeding practices, promote linkages with family planning services and support disclosure by HIV+ mothers to partners, male attendance and male HIV treatment. Mothers leave MSGs 6 months postnatally. Volunteer MSG coordinators contact defaulting mothers visits using cell phones; VHWs may conduct home visits to to defaulting MSG members to reduce LTFU;
  Interventions: Behavioral: Mother support groups for HIV+ mothers
- Standard of Care Arm (No Intervention): Standard of Care: Nurses may identify HIV+ mothers lost to follow-up (LTFU); village health workers (VHWs) may conduct home visits to reduce LTFU of HIV+ mothers. LTFU activities are not standardised throughout all Ministry of Health and Child Care facilities.

INTERVENTIONS:
Behavioral: Mother support groups for HIV+ mothers — Facility-based mother support groups (MSGs) for HIV+ mothers. MSGs were established prior to study enrolment. MSGs are facilitated by volunteer mothers. Groups meet every two weeks. Health information is provided by health workers during MSGs. Mothers receive HIV prevention, psychosocial and treatment support, reinforce safe feeding practices, promote linkages with family planning services and support disclosure by HIV+ mothers to partners, male attendance and male HIV treatment. Mothers leave MSGs 6 months postnatally. Volunteer MSG coordinators contact defaulting mothers visits using cell phones; VHWs may conduct home visits to to defaulting MSG members to reduce LTFU;
  Arms: Mother support groups for HIV+ mothers

SUMMARY:
The investigators hypothesize that a strategy of establishing facility-based mother support groups (MSGs) for HIV-positive mothers will result in increased retention rates of HIV-exposed infants in clinic-based PMTCT follow-up systems twelve months post-delivery compared to clinics that lack MSGs. The study will be conducted in health facilities in rural Mutare and Makoni health districts in Manicaland province, Zimbabwe. A two-arm cluster controlled study design will be used in 30 rural clinics randomly assigned to either arm to compare the effectiveness of MSGs. Arm 1 of the study consists of standard of care whilst arm 2 consists of standard of care together with facility-based MSGs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE To test whether MSGs lead to increased retention of HIV-exposed infants in PMTCT programmes

SECONDARY OBJECTIVES

1. To assess whether MSGs lead to increased retention of mothers in postnatal HIV follow-up care
2. To assess whether male participation in PMTCT activities is increased at clinics with MSGs
3. To assess whether selected maternal and infant health indicators are improved in HIV-positive mothers and their exposed infants at facilities with MSGs, viz. (1) Antenatal attendance; (2) Delivery in facilities; (3) Infant immunisation uptake; (4) Infant feeding methods and nutrition status; (5) Infant nevirapine prophylaxis; (6) Infant co-trimoxazole prophylaxis; (7) Infant HIV testing; and (8) Family planning uptake

MOTHER SUPPORT GROUP INTERVENTION MSGs were designed following formative research. A non-governmental organisation established MSGs by recruiting HIV+ mothers and volunteer coordinators (MSGCs) prior to commencing enrolment. MSGCs were HIV-positive mothers who were trained in MSG establishment and maintenance, retention activities and data collection. MSGs meet each two weeks with the MSGC or health worker facilitating an information session using a curriculum of eight PMTCT-related topics. MSGCs send standard message reminders to members, contact non-attending members by phone and inform health workers (HWs) to assist retention. HWs conduct retention actions of non-attending patients in PMTCT programmes.

SAMPLE SIZE AND RANDOMISATION We excluded from the study low-volume facilities that recorded booking fewer than 10 HIV-positive antenatal mothers per annum. We randomly selected facilities in the two study districts to either of the study arms. Based on estimated infant retention rates for control and intervention arms, we calculated the minimum sample size of 10 HIV-positive mothers to be enrolled at each health facility.

DATA COLLECTION, ANALYSIS AND QUALITY ASSURANCE The study utilizes the existing health information system (e.g. antenatal care (ANC) Register, Exposed Infant Follow-Up Register, Anti-retroviral treatment (ART) Register), supplemented by EPAZ study-related data collection and patient tracking systems. Study staff will work with clinic- and district-level staff to improve and collect routine and study-specific data. Data will be entered, coded, cleaned and locked before analyses are made. Data will be analysed on an intention-to-treat basis. A mobile team of well-trained quality assurance and control study staff will be deployed throughout the data collection period to ensure quality of the intervention and of data generated and collected at each study site. A pre-specified proportion of patient visit records will be reviewed from each site.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers
* with documented HIV-1 infection attending an antenatal clinic for the current pregnancy
* Aged 18 years of age or greater
* Attending the clinic with no known intention at the time of enrolment to permanently migrate outside the catchment area of the clinic for the duration of the study follow-up period
* Estimated gestational age of 34 weeks or less at time of enrolment
* Willing to have her infant, when born, participate in the study.
* Able and willing to give informed consent to participate

Exclusion Criteria:

* Pregnant mothers with no documented HIV infection
* Under 18 years of age
* Not able or willing to give informed consent to participate
* Estimated gestational age of over 34 weeks when considered for possible enrolment
* Not residing in catchment area of clinic
* Planning to relocate out of the catchment area of the clinic for the duration of study follow-up period or longer
* Any condition that in the opinion of the investigators would interfere with adherence to study requirements. Such conditions include mental illness or active drug or alcohol use or dependence.
* Unwilling for her infant, when born, to participate in the infant component of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
One-year retention rates of HIV-exposed infants in post-natal follow-up | 12 months postnatal

SECONDARY OUTCOMES:
a. Retention rates of HIV-infected mothers | 12 months postnatal

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Foster, MB BS MRCP, Principal Investigator — Ministry of Health and Child Welfare, Zimbabwe
Locations (1):
- Family AIDS Caring Trust, Mutare, Manicaland Province, Zimbabwe

REFERENCES:
- [Derived] Cataldo F, Sam-Agudu NA, Phiri S, Shumba B, Cornelius LJ, Foster G. The Roles of Expert Mothers Engaged in Prevention of Mother-to-Child Transmission (PMTCT) Programs: A Commentary on the INSPIRE Studies in Malawi, Nigeria, and Zimbabwe. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S224-S232. doi: 10.1097/QAI.0000000000001375. PMID 28498193
- [Derived] Foster G, Orne-Gliemann J, Font H, Kangwende A, Magezi V, Sengai T, Rusakaniko S, Shumba B, Zambezi P, Maphosa T. Impact of Facility-Based Mother Support Groups on Retention in Care and PMTCT Outcomes in Rural Zimbabwe: The EPAZ Cluster-Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S207-S215. doi: 10.1097/QAI.0000000000001360. PMID 28498191
- [Derived] Foster G, Kangwende A, Magezi V, Maphosa T, Mashapa R, Mukora-Mutseyekwa F, Mushavi A, Rusakaniko S, Shumba B, Zambezi P. Cluster randomized trial on the effect of mother support groups on retention-in-care and PMTCT outcomes in Zimbabwe: study design, challenges, and national relevance. J Acquir Immune Defic Syndr. 2014 Nov 1;67 Suppl 2:S145-9. doi: 10.1097/QAI.0000000000000325. PMID 25310121